CLINICAL TRIAL: NCT01293539
Title: Intra-arterial Chemotherapy for the Treatment of Intraocular Retinoblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IAC is now recognized as part of standard of care treatment options in the US.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1071; NA_00040637 (Other: JHMIRB)
Record Dates: First submitted 2011-01-21; First posted 2011-02-10 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; intra-arterial chemotherapy; angiography
MeSH Terms: conditions — Retinoblastoma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraocular Retinoblastoma Patients (Other): Single group assignment of patients with intraocular retinoblastoma, unilateral or bilateral.
  Interventions: Drug: Melphalan hydrochloride

INTERVENTIONS:
Drug: Melphalan hydrochloride — Drug administered intra-arterially (injection in the artery).
  Standard dose:
  2.5mg (3-6 month old) 3.0 mg (6-12 month old) 4.0 mg (1-3 year old) 5.0 mg (>3 years old)
  Dose modification: decrease standard dose by 25% if there are signs of toxicity. Increase the dose by 25% if there is inadequate tumor response.
  Frequency: 2 treatment cycles at 3-4 week intervals, with a third treatment cycle administered if the tumor requires it.
  Dose not to exceed 0.5mg/kg, per treatment cycle.
  Other Names: Alkeran

SUMMARY:
The purpose of this study is to show that chemotherapy delivered directly through the artery supplying the eye (ophthalmic artery) to patients with retinoblastoma is a safe and effective treatment alternative to conventional systemic chemotherapy, external beam radiation, and surgical removal of the eye.

DETAILED DESCRIPTION:
Delivering the chemotherapeutic agent in the arterial system through the ophthalmic artery transforms the treatment of retinoblastoma from systemic chemotherapy to local chemotherapy. Administration of the drug directly to the targeted site thus avoids the complications and adverse events associated with toxicity from systemic, rather than local, chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients newborn to 18 years old.
* Patients with intraocular retinoblastoma, unilateral or bilateral, who would be treated either by systemic chemotherapy, EBR, or enucleation would be considered for this study.

Exclusion Criteria:

* Patients over the age of 18.
* Patients with small, localized intraocular Rb amenable to focal therapy (laser or cryotherapy).
* Patients with extraocular disease evident on MRI (extension into the optic nerve), massive choroidal/uveal invasion (grade IIC or IID per ARET0332) or disease outside the globe evident on MRI or physical examination.
* Documented hypercoagulable disorders or vasculopathies.
* Laboratory exclusion criteria: GFR < 60 mL/min/1.73 m2

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Pearl, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Abramson DH, Dunkel IJ, Brodie SE, Kim JW, Gobin YP. A phase I/II study of direct intraarterial (ophthalmic artery) chemotherapy with melphalan for intraocular retinoblastoma initial results. Ophthalmology. 2008 Aug;115(8):1398-404, 1404.e1. doi: 10.1016/j.ophtha.2007.12.014. Epub 2008 Mar 14. PMID 18342944
- [Background] Abramson DH. Chemosurgery for retinoblastoma: what we know after 5 years. Arch Ophthalmol. 2011 Nov;129(11):1492-4. doi: 10.1001/archophthalmol.2011.354. No abstract available. PMID 22084221

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-arterial Chemotherapy: IAC is offered to all patients with intraocular Rb who are deemed eligible after evaluation under anesthesia (EUA),with the exception of those few patients for whom focal modalities (i.e., laser or cryotherapy) would be effective.In cases of bilateral disease, both eyes would be treated sequentially during the same procedure utilizing the same femoral access site.
  Two cycles of IAC will be performed at 3 to 4 week intervals. Melphalan dosing: 3-6 mth-old, 2.5mg; 3-12 mth-old, 3mg; 1-3 yr-old, 4mg; >3 yr-old, 5mg. For those tumors that have shown appropriate response and are amenable to local therapies, then no additional IAC will be performed. If the tumors do not regress after 2 cycles, then a third cycle of IAC will be offered. Local therapies (laser, cryotherapy) will not be given during the EUAs conducted prior to each treatment session, but will be allowed after toxicity and response has been assessed 3-4 weeks after the final cycle of intra-arterial therapy.
Period: Overall Study
Arm/Group | Intra-arterial Chemotherapy
Started | 10
Completed | 9
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intra-arterial Chemotherapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Complete Therapy Without the Need for Additional Treatment Including Systemic Chemotherapy, External Beam Radiation, or Enucleation.
Description: The primary objective of this study is to show that intra-arterial delivery of the chemotherapeutic agent is successful in treating intraocular retinoblastoma, defined as avoiding systemic chemotherapy, external beam radiation, and enucleation.
Time Frame: Within the first six months after the initial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-arterial Chemotherapy
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 4.5 years
Arm/Group | Intra-arterial Chemotherapy
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intra-arterial Chemotherapy (N=10)
Glaucoma (Eye disorders) | 2 (2) — Eye-disorder, Grade 1
Retinal vascular disorder (Eye disorders) | 1 (1) — Eye-disorder, Grade 2
Retinal vascular disorder (Eye disorders) | 1 (1) — Eye-disorder, Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intra-arterial Chemotherapy (N=10)
Eyelid edema & erythema (Eye disorders) | 1 (1) — Eyelid disorder, Grade 1
Eyelid function disorder (Eye disorders) | 1 (1) — Eye disorder, Grade 1
Injury - cut to lip during play (Injury, poisoning and procedural complications) | 1 (1) — Injury, Grade 2
Eyelid function disorder (Eye disorders) | 1 (1) — Eye disorder, Grade 2
Eye pain (Eye disorders) | 1 (1) — Eye disorder, Grade 1
Mild swelling (Eye disorders) | 1 (1) — Eye disorders, other, Grade 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Cough, Grade 1
Conjunctivitis (Eye disorders) | 1 (1) — Conjunctivitis, Grade 2
Flu-like symptoms (General disorders) | 1 (1) — Flu-like symptoms, Grade 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Cough, Grade 2
Vomiting (Gastrointestinal disorders) | 1 (1) — Vomiting, Grade 1
Fever (General disorders) | 1 (1) — Fever, Grade 2
Fever (General disorders) | 1 (1) — Fever, Grade 1
Ear infection (Infections and infestations) | 1 (1) — Otitis media, Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes